CLINICAL TRIAL: NCT02898454
Title: A Randomized, Double-blind, 52-week, Placebo Controlled Efficacy and Safety Study of Dupilumab, in Patients With Bilateral Nasal Polyposis on a Background Therapy With Intranasal Corticosteroids
Brief Title: Controlled Clinical Study of Dupilumab in Patients With Nasal Polyps
Acronym: SINUS-52
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EFC14280; 2015-001314-10 (EudraCT Number); U1111-1170-7180 (Other: UTN)
Record Dates: First submitted 2016-09-08; First posted 2016-09-13 (Estimated); Results first posted 2019-10-23 (Actual); Last update posted 2019-10-23 (Actual); Status verified 2019-10

CONDITIONS: Chronic Rhinosinusitis Phenotype With Nasal Polyps (CRSwNP)
MeSH Terms: interventions — dupilumab; Mometasone Furoate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Dupilumab 300 mg q2w (Experimental): Dupilumab 300 mg subcutaneous (SC) injection q2w from Day 1 of Week 0 up to Week 52 added to background therapy of intranasal MFNS at stable dose.
  Interventions: Drug: Dupilumab SAR231893 (REGN668); Drug: Mometasone furoate nasal spray
- Dupilumab 300 mg q2w then q4w (Experimental): Dupilumab 300 mg SC injection q2w from Day 1 of Week 0 up to Week 24 and then 300 mg q4w until Week 52 added to background therapy of intranasal MFNS at stable dose. After Week 24, Dupilumab administration was alternated with matched placebo injection every other week up to Week 50.
  Interventions: Drug: Dupilumab SAR231893 (REGN668); Drug: Placebo; Drug: Mometasone furoate nasal spray
- Placebo (Placebo Comparator): Placebo (for dupilumab), 1 SC injection q2w from Day 1 of Week 0 up to Week 52 added to background therapy of intranasal MFNS at stable dose.
  Interventions: Drug: Placebo; Drug: Mometasone furoate nasal spray

INTERVENTIONS:
Drug: Dupilumab SAR231893 (REGN668) — Pharmaceutical form: Solution
  Route of administration: Subcutaneous
  Arms: Dupilumab 300 mg q2w; Dupilumab 300 mg q2w then q4w
Drug: Placebo — Pharmaceutical form: Solution
  Route of administration: Subcutaneous
  Arms: Dupilumab 300 mg q2w then q4w; Placebo
Drug: Mometasone furoate nasal spray — Pharmaceutical form: Suspension
  Route of administration: Intranasal
  Other Names: NASONEX®

SUMMARY:
Primary Objective:

To evaluate the efficacy of dupilumab 300 mg every 2 weeks (q2w) compared to placebo on a background of mometasone furoate nasal spray (MFNS) in reducing nasal congestion (NC)/obstruction severity and endoscopic nasal polyp score (NPS) in participants with bilateral nasal polyps (NP). In addition for Japanese participants, reduction in computed tomography (CT) scan opacification of the sinuses was a co-primary objective.

Secondary Objectives:

* To evaluate the efficacy of dupilumab in improving total symptoms score.
* To evaluate the efficacy of dupilumab in improving sense of smell.
* To evaluate the efficacy of dupilumab in reducing CT scan opacification of the sinuses (primary objective for Japanese participants).
* To evaluate ability of dupilumab in reducing proportion of participants who required treatment with systemic corticosteroids (SCS) or surgery for NP.
* To evaluate the effect of dupilumab on participant reported outcomes and health related quality of life.
* To evaluate the efficacy of dupilumab 300 mg q2w up to Week 52.
* To evaluate the efficacy of dupilumab 300 mg q2w up to Week 24 followed by 300 mg every 4 weeks (q4w) up to Week 52.
* To evaluate the effect of dupilumab in the subgroups of participants with prior surgery and comorbid asthma including non-steroid anti-inflammatory drug exacerbated respiratory disease.
* To evaluate the safety of dupilumab in participants with bilateral NP.
* To evaluate functional dupilumab concentrations (systemic exposure) and incidence of treatment emergent anti-drug antibodies.

DETAILED DESCRIPTION:
The total study duration per participant was up to 68 weeks that consisted of a 4-weeks run-in period, 52-weeks treatment period, and a 12-weeks post treatment period.

ELIGIBILITY:
Inclusion criteria :

* Participants with bilateral sino-nasal polyposis that despite prior treatment with SCS anytime within the past 2 years; and/or had a medical contraindication/intolerance to SCS; and/or had prior surgery for NP at the screening visit, had:
* An endoscopic bilateral NPS at Visit 1 (V1) of at least 5 out of a maximum score of 8 (with a minimum score of 2 in each nasal cavity).
* Ongoing symptoms (for at least 8 weeks before V1) of NC/blockage/obstruction with moderate or severe symptom severity (score 2 or 3) at V1 and a weekly average severity of greater than 1 at time of randomization (V2), and another symptom such as loss of smell, rhinorrhea (anterior/posterior).
* Signed written informed consent.

Exclusion criteria:

* Participants <18 years of age.
* Participant who had been previously treated in dupilumab studies.
* Participant who had taken:

  * Biologic therapy/ systemic immunosuppressant to treat inflammatory disease or autoimmune disease (eg, rheumatoid arthritis, inflammatory bowel disease, primary biliary cirrhosis, systemic lupus erythematosus, multiple sclerosis, etc.) within 2 months before V1 or 5 half-lives, whichever was longer.
  * Any experimental monoclonal antibody within 5 half-lives or within 6 months before V1 if the half-life was unknown.
  * Anti-immunoglobulin E therapy (omalizumab) within 130 days prior to V1.
  * Participants who received leukotriene antagonists/modifiers at V1 unless they were on a continuous treatment for at least 30 days prior to V1.
* Initiation of allergen immunotherapy within 3 months prior to V1 or a plan to begin therapy or change its dose during the run-in period or the randomized treatment period.
* Participants who underwent any and/or sinus surgery (including polypectomy) within 6 months before V1.
* Participants who had a sino-nasal or sinus surgery changing the lateral wall structure of the nose making impossible the evaluation of NPS.
* Participants with conditions/concomitant diseases making them non evaluable at V1 or for the primary efficacy endpoint such as:

  * Antrochoanal polyps,
  * Nasal septal deviation that would occlude at least one nostril,
  * Acute sinusitis, nasal infection or upper respiratory infection,
  * Ongoing rhinitis medicamentosa,
  * Allergic granulomatous angiitis (Churg-Strauss syndrome), granulomatosis with polyangiitis (Wegener's granulomatosis),Young's syndrome, Kartagener's syndrome or other dyskinetic ciliary syndromes, concomitant cystic fibrosis,
  * Radiologic suspicion, or confirmed invasive or expansive fungal rhinosinusitis.
* Participants with nasal cavity malignant tumor and benign tumors (eg, papilloma, blood boil etc.).
* Participants with forced expiratory volume 50% or less (of predicted normal).
* Participants who received concomitant treatment prohibited in the study.
* Treatment with a live (attenuated) vaccine within 4 weeks before the baseline visit.
* Treatment with a live (attenuated) vaccine within 12 weeks before the baseline visit.
* History of human immunodeficiency virus (HIV) infection or positive HIV serology at screening.
* Positive with hepatitis B surface antigen or hepatitis C antibody at the screening visit.
* Active chronic or acute infection requiring systemic treatment within 2 weeks before the baseline visit.
* Known or suspected history of immunosuppression.
* Pregnant or breastfeeding women, or women planning to become pregnant or breastfeed during the study.
* Women unwilling to use adequate birth control, if of reproductive potential and sexually active.

The above information was not intended to contain all considerations relevant to a Participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 448 (Actual)
Dates: Start 2016-11-28 (Actual); Primary Completion 2018-08-27 (Actual); Study Completion 2018-11-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (123):
- United States (19):
  - Investigational Site Number 8400019, Birmingham, Alabama
  - Investigational Site Number 8400011, Fresno, California
  - Investigational Site Number 8400008, Huntington Beach, California
  - Investigational Site Number 8400004, Rolling Hills Estates, California
  - Investigational Site Number 8400012, Walnut Creek, California
  - Investigational Site Number 8400017, Colorado Springs, Colorado
  - Investigational Site Number 8400006, Denver, Colorado
  - Investigational Site Number 8400022, New Haven, Connecticut
  - Investigational Site Number 8400002, Louisville, Kentucky
  - Investigational Site Number 8400021, Boston, Massachusetts
  - Investigational Site Number 8400014, Kansas City, Missouri
  - Investigational Site Number 8400024, The Bronx, New York
  - Investigational Site Number 8400016, North Charleston, North Carolina
  - Investigational Site Number 8400013, Bethlehem, Pennsylvania
  - Investigational Site Number 8400005, Philadelphia, Pennsylvania
  - Investigational Site Number 8400003, Pittsburgh, Pennsylvania
  - Investigational Site Number 8400009, Salt Lake City, Utah
  - Investigational Site Number 8400010, Bellevue, Washington
  - Investigational Site Number 8400007, Milwaukee, Wisconsin
- Argentina (8):
  - Investigational Site Number 0320006, Buenos Aires
  - Investigational Site Number 0320004, Buenos Aires
  - Investigational Site Number 0320005, Caba
  - Investigational Site Number 0320001, Caba
  - Investigational Site Number 0320007, Caba
  - Investigational Site Number 0320003, Mendoza
  - Investigational Site Number 0320008, Rosario
  - Investigational Site Number 0320002, San Miguel de Tucumán
- Australia (5):
  - Investigational Site Number 0360002, Clayton
  - Investigational Site Number 0360004, Herston
  - Investigational Site Number 0360005, Murdoch
  - Investigational Site Number 0360001, Parkville
  - Investigational Site Number 0360003, Prahran
- Belgium (3):
  - Investigational Site Number 0560003, Brussels
  - Investigational Site Number 0560001, Ghent
  - Investigational Site Number 0560002, Leuven
- Canada (8):
  - Investigational Site Number 1240007, Kingston
  - Investigational Site Number 1240002, Montreal
  - Investigational Site Number 1240006, Montreal
  - Investigational Site Number 1240005, Ottawa
  - Investigational Site Number 1240003, Québec
  - Investigational Site Number 1240004, Québec
  - Investigational Site Number 1240008, Trois-Rivières
  - Investigational Site Number 1240001, Vancouver
- Chile (10):
  - Investigational Site Number 1520009, Quillota
  - Investigational Site Number 1520010, San Fernando
  - Investigational Site Number 1520005, Santiago
  - Investigational Site Number 1520011, Santiago
  - Investigational Site Number 1520008, Santiago
  - Investigational Site Number 1520006, Santiago
  - Investigational Site Number 1520001, Santiago
  - Investigational Site Number 1520014, Santiago
  - Investigational Site Number 1520003, Talca
  - Investigational Site Number 1520007, Viña del Mar
- Israel (5):
  - Investigational Site Number 3760001, Hadera
  - Investigational Site Number 3760003, Nahariya
  - Investigational Site Number 3760002, Petah Tikva
  - Investigational Site Number 3760005, Rehovot
  - Investigational Site Number 3760004, Tel Litwinsky
- Japan (29):
  - Investigational Site Number 3920004, Bunkyō City
  - Investigational Site Number 3920009, Bunkyō City
  - Investigational Site Number 3920026, Bunkyō City
  - Investigational Site Number 3920006, Chiyoda-Ku
  - Investigational Site Number 3920024, Fukuoka
  - Investigational Site Number 3920010, Hirakata-Shi
  - Investigational Site Number 3920011, Hiroshima
  - Investigational Site Number 3920007, Iida-Shi
  - Investigational Site Number 3920015, Inzai-Shi
  - Investigational Site Number 3920012, Itabashi-Ku
  - Investigational Site Number 3920014, Izumisano
  - Investigational Site Number 3920016, Kawasaki-Shi
  - Investigational Site Number 3920020, Kitakyushu-Shi
  - Investigational Site Number 3920027, Kitakyushu-Shi
  - Investigational Site Number 3920002, Kumamoto
  - Investigational Site Number 3920021, Kumamoto
  - Investigational Site Number 3920003, Kyoto
  - Investigational Site Number 3920023, Meguro-Ku
  - Investigational Site Number 3920013, Moriguchi-Shi
  - Investigational Site Number 3920025, Okayama
  - Investigational Site Number 3920018, Osaka
  - Investigational Site Number 3920017, Ōta-ku
  - Investigational Site Number 3920005, Sendai
  - Investigational Site Number 3920022, Sendai
  - Investigational Site Number 3920001, Shimonoseki-Shi
  - Investigational Site Number 3920029, Shinagawa-Ku
  - Investigational Site Number 3920030, Shinjyuku-Ku
  - Investigational Site Number 3920028, Takatsuki-Shi
  - Investigational Site Number 3920019, Yoshida-Gun
- Mexico (5):
  - Investigational Site Number 4840001, Chihuahua City
  - Investigational Site Number 4840005, Chihuahua City
  - Investigational Site Number 4840004, Durango
  - Investigational Site Number 4840002, Guadalajara
  - Investigational Site Number 4840003, Monterrey
- Portugal (6):
  - Investigational Site Number 6200004, Aveiro
  - Investigational Site Number 6200006, Guimarães
  - Investigational Site Number 6200002, Lisbon
  - Investigational Site Number 6200007, Matosinhos Municipality
  - Investigational Site Number 6200001, Porto
  - Investigational Site Number 6200005, Viana do Castelo
- Russia (5):
  - Investigational Site Number 6430006, Moscow
  - Investigational Site Number 6430003, Odintsovo
  - Investigational Site Number 6430002, Saint Petersburg
  - Investigational Site Number 6430005, Stavropol
  - Investigational Site Number 6430001, Yaroslavl
- Spain (6):
  - Investigational Site Number 7240001, Barcelona
  - Investigational Site Number 7240006, Barcelona
  - Investigational Site Number 7240003, Jerez de la Frontera
  - Investigational Site Number 7240002, Madrid
  - Investigational Site Number 7240007, Seville
  - Investigational Site Number 7240009, Valencia
- Sweden (2):
  - Investigational Site Number 7520002, Lund
  - Investigational Site Number 7520001, Stockholm
- Turkey (Türkiye) (12):
  - Investigational Site Number 7920004, Ankara
  - Investigational Site Number 7920005, Ankara
  - Investigational Site Number 7920008, Ankara
  - Investigational Site Number 7920013, Bursa
  - Investigational Site Number 7920010, Istanbul
  - Investigational Site Number 7920009, Istanbul
  - Investigational Site Number 7920003, Istanbul
  - Investigational Site Number 7920001, Istanbul
  - Investigational Site Number 7920002, Istanbul
  - Investigational Site Number 7920006, Izmir
  - Investigational Site Number 7920007, Izmir
  - Investigational Site Number 7920011, Rize

IPD SHARING:
Plan to Share IPD: No
Not available for request

REFERENCES:
- [Derived] Bachert C, Khan AH, Hopkins C, Han JK, Fokkens WJ, Mannent LP, Msihid J, Borsos K, Kamat S, Nash S, Sacks H, Rowe PJ, Deniz Y, Jacob-Nara JA. Mild and symptom-free months in patients with chronic rhinosinusitis with nasal polyps treated with dupilumab. Ann Allergy Asthma Immunol. 2025 Jan;134(1):61-69.e12. doi: 10.1016/j.anai.2024.09.015. Epub 2024 Sep 28. PMID 39343385
- [Derived] Bachert C, Khan AH, Fokkens WJ, Hopkins C, Gevaert P, Han JK, Hellings PW, Lee SE, Msihid J, Nash S, Sacks H, Jacob-Nara JA, Deniz Y, Rowe PJ. Dupilumab response onset, maintenance, and durability in patients with severe CRSwNP. J Allergy Clin Immunol. 2024 Dec;154(6):1442-1449. doi: 10.1016/j.jaci.2024.07.026. Epub 2024 Aug 14. PMID 39151476
- [Derived] Fokkens WJ, Bachert C, Hopkins C, Marglani O, Praestgaard A, Nash S, Deniz Y, Rowe PJ, Sacks H, Jacob-Nara JA. Dupilumab improves outcomes in patients with chronic rhinosinusitis with nasal polyps irrespective of gender: results from the SINUS-52 trial. Clin Transl Immunology. 2024 Jun 8;13(6):e1511. doi: 10.1002/cti2.1511. eCollection 2024. PMID 38854740
- [Derived] Hopkins C, Mullol J, Khan AH, Lee SE, Wagenmann M, Hellings P, Fokkens W, Msihid J, Nair R, Kamat S, Nash S, Radwan A, Jacob-Nara JA, Deniz Y, Rowe PJ. Impact of Dupilumab on Sinonasal Symptoms and Outcomes in Severe Chronic Rhinosinusitis With Nasal Polyps. Otolaryngol Head Neck Surg. 2024 Apr;170(4):1173-1182. doi: 10.1002/ohn.627. Epub 2023 Dec 29. PMID 38156522
- [Derived] Lee SE, Amin N, Mannent LP, Bachert C, Gross G, Cho SH, Praestgaard A, Siddiqui S, Nash S, Kamat S, Khan AH, Jacob Nara JA. The relationship of sinus opacification, olfaction and dupilumab efficacy in patients with CRSwNP. Rhinology. 2023 Dec 1;61(6):531-540. doi: 10.4193/Rhin22.220. PMID 37453138
- [Derived] Bachert C, Laidlaw TM, Cho SH, Mullol J, Swanson BN, Naimi S, Classe M, Harel S, Jagerschmidt A, Laws E, Ruddy M, Praestgaard A, Amin N, Mannent LP. Effect of Dupilumab on Type 2 Biomarkers in Chronic Rhinosinusitis With Nasal Polyps: SINUS-52 Study Results. Ann Otol Rhinol Laryngol. 2023 Dec;132(12):1649-1661. doi: 10.1177/00034894231176334. Epub 2023 Jun 15. PMID 37322842
- [Derived] Maspero JF, Bachert C, Martinez FJ, Hanania NA, Ortiz B, Patel N, Mannent LP, Praestgaard A, Pandit-Abid N, Siddiqui S, Hardin M. Clinical Efficacy among Patients with Chronic Rhinosinusitis with Nasal Polyps and Clinical Features of Obstructive Lung Disease: Post Hoc Analysis of the Phase III SINUS-24 and SINUS-52 Studies. J Asthma Allergy. 2023 Mar 31;16:333-342. doi: 10.2147/JAA.S357393. eCollection 2023. PMID 37026112
- [Derived] Gevaert P, Lee SE, Settipane RA, Wagenmann M, Msihid J, Siddiqui S, Nash S, Jacob-Nara JA, Khan AH, Kamat S, Chuang CC. Dupilumab provides early and durable improvement of symptoms in patients with chronic rhinosinusitis with nasal polyps. Clin Transl Immunology. 2023 Jan 27;12(1):e1433. doi: 10.1002/cti2.1433. eCollection 2023. PMID 36721661
- [Derived] Peters AT, Soler ZM, Kern RC, Heffler E, Maspero JF, Crampette L, Fujieda S, Lane AP, Zhang H, Nash S, Khan AH, Siddiqui S, Jacob-Nara JA, Rowe P, Deniz Y. Improvement in patient-reported "taste" and association with smell in dupilumab-treated patients with severe chronic rhinosinusitis with nasal polyps from the SINUS-24 and SINUS-52 trials. Clin Exp Allergy. 2022 Sep;52(9):1105-1109. doi: 10.1111/cea.14194. Epub 2022 Jul 12. No abstract available. PMID 35775319
- [Derived] Wechsler ME, Klion AD, Paggiaro P, Nair P, Staumont-Salle D, Radwan A, Johnson RR, Kapoor U, Khokhar FA, Daizadeh N, Chen Z, Laws E, Ortiz B, Jacob-Nara JA, Mannent LP, Rowe PJ, Deniz Y. Effect of Dupilumab on Blood Eosinophil Counts in Patients With Asthma, Chronic Rhinosinusitis With Nasal Polyps, Atopic Dermatitis, or Eosinophilic Esophagitis. J Allergy Clin Immunol Pract. 2022 Oct;10(10):2695-2709. doi: 10.1016/j.jaip.2022.05.019. Epub 2022 May 28. PMID 35636689
- [Derived] Bachert C, Peters AT, Heffler E, Han JK, Olze H, Pfaar O, Chuang CC, Rout R, Attre R, Goga L, Jacob-Nara JA, Rowe PJ, Deniz Y, Chen Z, Kamat S, Siddiqui S. Responder analysis to demonstrate the effect of targeting type 2 inflammatory mechanisms with dupilumab across objective and patient-reported endpoints for patients with severe chronic rhinosinusitis with nasal polyps in the SINUS-24 and SINUS-52 studies. Clin Exp Allergy. 2022 Feb;52(2):244-249. doi: 10.1111/cea.14051. No abstract available. PMID 35092110
- [Derived] Lee SE, Hopkins C, Mullol J, Msihid J, Guillemin I, Amin N, Mannent LP, Li Y, Siddiqui S, Chuang CC, Kamat S, Khan AH. Dupilumab improves health related quality of life: Results from the phase 3 SINUS studies. Allergy. 2022 Jul;77(7):2211-2221. doi: 10.1111/all.15222. Epub 2022 Feb 1. PMID 35034364
- [Derived] Bachert C, Corren J, Lee SE, Zhang H, Harel S, Cunoosamy D, Khan AH, Jacob-Nara JA, Siddiqui S, Nash S, Rowe PJ, Deniz Y. Dupilumab efficacy and biomarkers in chronic rhinosinusitis with nasal polyps: Association between dupilumab treatment effect on nasal polyp score and biomarkers of type 2 inflammation in patients with chronic rhinosinusitis with nasal polyps in the phase 3 SINUS-24 and SINUS-52 trials. Int Forum Allergy Rhinol. 2022 Sep;12(9):1191-1195. doi: 10.1002/alr.22964. Epub 2022 Jan 31. No abstract available. PMID 34970860
- [Derived] Geng B, Bachert C, Busse WW, Gevaert P, Lee SE, Niederman MS, Chen Z, Lu X, Khokhar FA, Kapoor U, Pandit-Abid N, Jacob-Nara JA, Rowe PJ, Deniz Y, Ortiz B. Respiratory Infections and Anti-Infective Medication Use From Phase 3 Dupilumab Respiratory Studies. J Allergy Clin Immunol Pract. 2022 Mar;10(3):732-741. doi: 10.1016/j.jaip.2021.12.006. Epub 2021 Dec 22. PMID 34954123
- [Derived] Hellings PW, Peters AT, Chaker AM, Heffler E, Zhang H, Praestgaard A, Nash S, Khan AH, Siddiqui S, Jacob-Nara JA, Rowe PJ, Deniz Y. Rapid and sustained effects of dupilumab in severe chronic rhinosinusitis with nasal polyps. Int Forum Allergy Rhinol. 2022 Jul;12(7):958-962. doi: 10.1002/alr.22944. Epub 2022 Jan 23. No abstract available. PMID 34911163
- [Derived] Han JK, Bachert C, Lee SE, Hopkins C, Heffler E, Hellings PW, Peters AT, Kamat S, Whalley D, Qin S, Nelson L, Siddiqui S, Khan AH, Li Y, Mannent LP, Guillemin I, Chuang CC. Estimating Clinically Meaningful Change of Efficacy Outcomes in Inadequately Controlled Chronic Rhinosinusitis with Nasal Polyposis. Laryngoscope. 2022 Feb;132(2):265-271. doi: 10.1002/lary.29888. Epub 2021 Dec 1. PMID 34850966
- [Derived] Chuang CC, Guillemin I, Bachert C, Lee SE, Hellings PW, Fokkens WJ, Duverger N, Fan C, Daizadeh N, Amin N, Mannent LP, Khan AH, Kamat S. Dupilumab in CRSwNP: Responder Analysis Using Clinically Meaningful Efficacy Outcome Thresholds. Laryngoscope. 2022 Feb;132(2):259-264. doi: 10.1002/lary.29911. Epub 2021 Nov 24. PMID 34817082
- [Derived] Mullol J, Laidlaw TM, Bachert C, Mannent LP, Canonica GW, Han JK, Maspero JF, Picado C, Daizadeh N, Ortiz B, Li Y, Ruddy M, Laws E, Amin N. Efficacy and safety of dupilumab in patients with uncontrolled severe chronic rhinosinusitis with nasal polyps and a clinical diagnosis of NSAID-ERD: Results from two randomized placebo-controlled phase 3 trials. Allergy. 2022 Apr;77(4):1231-1244. doi: 10.1111/all.15067. Epub 2021 Oct 1. PMID 34459002
- [Derived] Khan AH, Reaney M, Guillemin I, Nelson L, Qin S, Kamat S, Mannent L, Amin N, Whalley D, Hopkins C. Development of Sinonasal Outcome Test (SNOT-22) Domains in Chronic Rhinosinusitis With Nasal Polyps. Laryngoscope. 2022 May;132(5):933-941. doi: 10.1002/lary.29766. Epub 2021 Aug 26. PMID 34437720
- [Derived] Hamilton JD, Harel S, Swanson BN, Brian W, Chen Z, Rice MS, Amin N, Ardeleanu M, Radin A, Shumel B, Ruddy M, Patel N, Pirozzi G, Mannent L, Graham NMH. Dupilumab suppresses type 2 inflammatory biomarkers across multiple atopic, allergic diseases. Clin Exp Allergy. 2021 Jul;51(7):915-931. doi: 10.1111/cea.13954. Epub 2021 Jun 26. PMID 34037993
- [Derived] Fujieda S, Matsune S, Takeno S, Ohta N, Asako M, Bachert C, Inoue T, Takahashi Y, Fujita H, Deniz Y, Rowe P, Ortiz B, Li Y, Mannent LP. Dupilumab efficacy in chronic rhinosinusitis with nasal polyps from SINUS-52 is unaffected by eosinophilic status. Allergy. 2022 Jan;77(1):186-196. doi: 10.1111/all.14906. Epub 2021 Jun 4. PMID 33993501
- [Derived] Chong LY, Piromchai P, Sharp S, Snidvongs K, Webster KE, Philpott C, Hopkins C, Burton MJ. Biologics for chronic rhinosinusitis. Cochrane Database Syst Rev. 2021 Mar 12;3(3):CD013513. doi: 10.1002/14651858.CD013513.pub3. PMID 33710614
- [Derived] Hopkins C, Wagenmann M, Bachert C, Desrosiers M, Han JK, Hellings PW, Lee SE, Msihid J, Radwan A, Rowe P, Amin N, Deniz Y, Ortiz B, Mannent LP, Rout R. Efficacy of dupilumab in patients with a history of prior sinus surgery for chronic rhinosinusitis with nasal polyps. Int Forum Allergy Rhinol. 2021 Jul;11(7):1087-1101. doi: 10.1002/alr.22780. Epub 2021 Feb 21. PMID 33611847
- [Derived] Peters AT, Han JK, Hellings P, Heffler E, Gevaert P, Bachert C, Xu Y, Chuang CC, Neupane B, Msihid J, Mannent LP, Guyot P, Kamat S. Indirect Treatment Comparison of Biologics in Chronic Rhinosinusitis with Nasal Polyps. J Allergy Clin Immunol Pract. 2021 Jun;9(6):2461-2471.e5. doi: 10.1016/j.jaip.2021.01.031. Epub 2021 Feb 4. PMID 33548517
- [Derived] Laidlaw TM, Bachert C, Amin N, Desrosiers M, Hellings PW, Mullol J, Maspero JF, Gevaert P, Zhang M, Mao X, Khan AH, Kamat S, Patel N, Graham NMH, Ruddy M, Staudinger H, Mannent LP. Dupilumab improves upper and lower airway disease control in chronic rhinosinusitis with nasal polyps and asthma. Ann Allergy Asthma Immunol. 2021 May;126(5):584-592.e1. doi: 10.1016/j.anai.2021.01.012. Epub 2021 Jan 16. PMID 33465455
- [Derived] Fujieda S, Matsune S, Takeno S, Asako M, Takeuchi M, Fujita H, Takahashi Y, Amin N, Deniz Y, Rowe P, Mannent L. The Effect of Dupilumab on Intractable Chronic Rhinosinusitis with Nasal Polyps in Japan. Laryngoscope. 2021 Jun;131(6):E1770-E1777. doi: 10.1002/lary.29230. Epub 2020 Nov 23. PMID 33226139
- [Derived] Bachert C, Han JK, Desrosiers M, Hellings PW, Amin N, Lee SE, Mullol J, Greos LS, Bosso JV, Laidlaw TM, Cervin AU, Maspero JF, Hopkins C, Olze H, Canonica GW, Paggiaro P, Cho SH, Fokkens WJ, Fujieda S, Zhang M, Lu X, Fan C, Draikiwicz S, Kamat SA, Khan A, Pirozzi G, Patel N, Graham NMH, Ruddy M, Staudinger H, Weinreich D, Stahl N, Yancopoulos GD, Mannent LP. Efficacy and safety of dupilumab in patients with severe chronic rhinosinusitis with nasal polyps (LIBERTY NP SINUS-24 and LIBERTY NP SINUS-52): results from two multicentre, randomised, double-blind, placebo-controlled, parallel-group phase 3 trials. Lancet. 2019 Nov 2;394(10209):1638-1650. doi: 10.1016/S0140-6736(19)31881-1. Epub 2019 Sep 19. PMID 31543428

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were involved in the study from 28 November 2016 to 16 November 2018 at 117 centers in 14 countries. A total of 806 participants were screened, of which 448 participants were enrolled and randomized to receive dupilumab 300 mg or placebo. A total of 358 participants had screen failures due to failure to meet inclusion criteria.
Pre-assignment Details: Randomization was stratified according to asthma and/or non-steroidal anti-inflammatory drug exacerbated respiratory disease (NSAID-ERD) history (yes/no), prior nasal polyps (NP) surgery (yes or not), and country.
Groups:
- Placebo: Placebo (for dupilumab), 1 subcutaneous (SC) injection every 2 weeks (q2w) from Day 1 of Week 0 up to Week 52 added to background therapy of intranasal mometasone furoate nasal spray (MFNS) at stable dose.
- Dupilumab 300 mg q2w Then q4w: Dupilumab 300 mg SC injection q2w from Day 1 of Week 0 up to Week 24 and then 300 mg every 4 weeks (q4w) until Week 52 added to background therapy of intranasal MFNS at stable dose. After Week 24, Dupilumab administration was alternated with matched placebo injection every other week up to Week 50.
- Dupilumab 300 mg q2w: Dupilumab 300 mg SC injection q2w from Day 1 of Week 0 up to Week 52 added to background therapy of intranasal MFNS at stable dose.
Period: Overall Study
Arm/Group | Placebo | Dupilumab 300 mg q2w Then q4w | Dupilumab 300 mg q2w
Started (Randomized population) | 153 | 145 | 150
Intent-to-Treat (ITT) Population (Randomized participants who were analyzed according to treatment group allocated by randomization.) | 153 | 145 | 150
Treated | 152 | 145 | 150
Safety Population | 150 (2 participants randomized to placebo received 1 dose of dupilumab:counted in 300 mg q2w then q4w arm) | 148 (1 randomized to dupilumab q2w arm received 1dose of placebo: counted in 300 mg q2w then q4w arm.) | 149
Completed | 136 | 140 | 144
Not Completed | 17 | 5 | 6
Not completed — Adverse Event | 4 | 1 | 2
Not completed — Protocol Violation | 1 | 0 | 1
Not completed — Lack of Efficacy | 4 | 1 | 0
Not completed — Withdrawal by Subject | 6 | 3 | 3
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Did Not Met Eligibility Criteria | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was performed on randomized population which included any participant who was allocated to a randomized treatment regardless of whether any treatment kit was used.
Groups:
- Dupilumab 300mg q2w: Dupilumab 300 mg SC injection q2w from Day 1 of Week 0 up to Week 52 added to background therapy of intranasal MFNS at stable dose.
- Total: Total of all reporting groups
Arm/Group | Placebo | Dupilumab 300 mg q2w Then q4w | Dupilumab 300mg q2w | Total
Number analyzed (Participants) | 153 | 145 | 150 | 448
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.67 (12.66) | 52.28 (12.87) | 51.91 (11.88) | 51.95 (12.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 58 | 53 | 169
  Male | 95 | 87 | 97 | 279
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 40 | 42 | 50 | 132
  Not Hispanic or Latino | 113 | 102 | 100 | 315
  Unknown or Not Reported | 0 | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian/White | 128 | 120 | 124 | 372
  Black/of African descent | 3 | 2 | 2 | 7
  Asian/Oriental | 18 | 19 | 17 | 54
  American Indian or Alaska Native | 3 | 2 | 7 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Multiple | 1 | 1 | 0 | 2
Nasal Congestion/Obstruction (NC) Symptom Severity Score [Mean (Standard Deviation); unit: score on a scale] — NC symptom severity was assessed by the participants on a scale of 0 to 3, where 0 = no symptoms, 1 = mild symptoms, 2 = moderate symptoms and 3 = severe symptoms, with higher scores indicated more severity.
  score on a scale | 2.38 (0.54) | 2.44 (0.59) | 2.48 (0.62) | 2.43 (0.59)
Nasal Polyp Score (NPS) [Mean (Standard Deviation); unit: score on a scale] — NPS was the sum of right and left nostril scores, as evaluated by means of nasal endoscopy. For each nostril, NPS was graded based on polyp size from 0 to 4 (0 = no polyps to 4 = large polyps causing complete obstruction of the inferior nasal cavity), with a lower score indicating smaller-sized polyps. Total NPS was the sum of right and left nostril scores and ranges from 0 (no polyps) to 8 (large polyps), with higher score representing more severe disease. Population: "Number analyzed" = Number of participants evaluable for the specified baseline measure.
  score on a scale
    number analyzed (Participants) | 152 | 145 | 149 | 446
    (all) | 5.96 (1.21) | 6.29 (1.20) | 6.07 (1.22) | 6.10 (1.21)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline at Week 24 in Nasal Congestion/Obstruction Symptom Severity Score
Description: NC symptom severity was assessed by the participants on a daily basis from visit 1 and throughout the study using an e-diary on a scale of 0 to 3, where 0 = no symptoms, 1 = mild symptoms, 2 = moderate symptoms and 3 = severe symptoms, with higher scores indicated more severity. Least squares (LS) means and standard error (SE) were obtained from Analysis of covariance (ANCOVA) model described in Statistical Analysis Overview. All participants randomized to receive Dupilumab had been on 300 mg q2w regimen until Week 24 and analyzed as a pooled population for Week 24 assessments.
Time Frame: Baseline, Week 24
Population: The analysis was performed on intent-to-treat (ITT) population which included all randomized participants who were analyzed according to the treatment group allocated by randomization. Data for this outcome measure was planned to be analyzed for the combined population of participants who received Dupilumab.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- Dupilumab 300 mg (24 Weeks Pooled Arm): Pooled arm consisted of all participants from both dupilumab treatment arms up to 24 weeks as both arms to this time point used the 300 mg q2w regimen.
Arm/Group | Placebo | Dupilumab 300 mg (24 Weeks Pooled Arm)
Number analyzed (Participants) | 153 | 295
score on a scale | -0.38 (0.07) | -1.25 (0.06)
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 300 mg (24 Weeks Pooled Arm); Data was analyzed using a hybrid method of the worst-observation carried forward (WOCF) and multiple imputation (MI). The imputed completed data were analyzed by fitting ANCOVA model with the corresponding baseline, treatment group, asthma/NSAID-ERD status, prior surgery history, and regions as covariates. Statistical inference obtained from all imputed data was combined using Rubin's rule; Test type: Superiority; p < 0.0001, ANCOVA; LS mean difference = -0.87, 95% CI 2-sided [-1.03 to -0.71]

2. Primary Outcome: Change From Baseline at Week 24 in Nasal Polyp Score
Description: NPS: sum of right, left nostril scores, evaluated by nasal endoscopy. For each nostril, NPS was graded based on polyp size from 0 = no polyps to 4 = large polyps causing complete obstruction of inferior nasal cavity; lower score = smaller sized polyps. Total NPS: sum of right and left nostril scores, ranges from 0 (no polyps) to 8 (large polyps), higher score = more severe disease. NPS was assessed by centralized, blinded, independent review of the nasal endoscopy video recordings. LS means and SE were obtained from ANCOVA model described in Statistical Analysis Overview. All participants randomized to receive Dupilumab had been on 300 mg q2w regimen until Week 24 and analyzed as a pooled population for Week 24 assessments.
Time Frame: Baseline, Week 24
Population: Analysis was performed on ITT population. Here, 'overall number of participants analyzed' = participants evaluable for this outcome measure. Data for this outcome measure was planned to be analyzed for the combined population of participants who received Dupilumab.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab 300 mg (24 Weeks Pooled Arm)
Number analyzed (Participants) | 152 | 294
score on a scale | 0.10 (0.14) | -1.71 (0.11)
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 300 mg (24 Weeks Pooled Arm); Data was analyzed using a hybrid method of the WOCF and MI. The imputed completed data were analyzed by fitting an ANCOVA model with corresponding baseline value, treatment group, asthma/NSAID-ERD status, prior surgery history, and regions as covariates. Statistical inference obtained from all imputed data was combined using Rubin's rule; Test type: Superiority; p < 0.0001, ANCOVA; LS mean difference = -1.80, 95% CI 2-sided [-2.10 to -1.51]

3. Secondary Outcome: Change From Baseline at Week 24 in Opacification of Sinuses Measured by Lund Mackay (LMK) Score
Description: The LMK scoring system rated each of both the left and right frontal, maxillary, sphenoid, ostiomeatal complex, anterior ethmoid and posterior ethmoid sinuses using following grading: 0 = normal, 1 = partial opacification, 2 = total opacification. The total score was the sum of scores from each side and ranges from 0 (normal) to 24 (more opacified); higher score indicated more severe disease. LS means and SE were obtained from ANCOVA model described in Statistical Analysis Overview. NOTE: For Japan regulatory submission only, this endpoint is not included as a secondary outcome measure and is instead one of the co-primary outcome measures. All participants randomized to receive Dupilumab had been on 300 mg q2w regimen until Week 24 and analyzed as a pooled population for Week 24 assessments.
Time Frame: Baseline, Week 24
Population: Analysis was performed on ITT population. Here, 'overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab 300 mg (24 Weeks Pooled Arm)
Number analyzed (Participants) | 150 | 289
score on a scale | -0.09 (0.31) | -5.21 (0.24)
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 300 mg (24 Weeks Pooled Arm); Data were analyzed using a hybrid method of the WOCF and MI. The imputed completed data were analyzed by fitting an ANCOVA model with corresponding baseline, treatment group, asthma/NSAID-ERD status, prior surgery history, and regions as covariates. Statistical inference obtained from all imputed data was combined using Rubin's rule; Test type: Superiority — Hierarchical testing procedure was used to control type I error. For regions outside of Japan, this first secondary endpoint was not tested unless both co-primary endpoints were significant at the 0.05 level. Hierarchical testing continued only when previous endpoint was statistically significant. For Japan submission, LMK was instead a co-primary endpoint which also had to be met before secondary endpoints were tested in the hierarchy. Last endpoint in hierarchy is Week 52 SNOT-22; p < 0.0001, ANCOVA — Threshold for significance at 0.05 level; LS mean difference = -5.13, 95% CI 2-sided [-5.80 to -4.46]

4. Secondary Outcome: Change From Baseline at Week 24 in Total Symptom Score (TSS)
Description: The TSS was the sum of participant-assessed nasal symptom scores for NC/obstruction, decreased/loss of sense of smell, and rhinorrhea (anterior/posterior nasal discharge), each accessed on 0-3 categorical scale (where 0 = no symptoms, 1 = mild symptoms, 2 = moderate symptoms and 3 = severe symptoms). Total score ranged from 0 (no symptoms) to 9 (severe symptoms). Higher score indicated more severe symptoms. LS means and SE were obtained from ANCOVA model described in Statistical Analysis Overview. All participants randomized to receive Dupilumab had been on 300 mg q2w regimen until Week 24 and analyzed as a pooled population for Week 24 assessments.
Time Frame: Baseline, Week 24
Population: Analysis was performed on ITT population. Data for this outcome measure was planned to be analyzed for the combined population of participants who received Dupilumab.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab 300 mg (24 Weeks Pooled Arm)
Number analyzed (Participants) | 153 | 295
score on a scale | -1.00 (0.20) | -3.45 (0.15)
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 300 mg (24 Weeks Pooled Arm); Data were analyzed using a hybrid method of the WOCF and MI. The imputed completed data were analyzed by fitting an ANCOVA model with corresponding baseline value, treatment group, asthma/NSAID-ERD status, prior surgery history, and regions as covariates. Statistical inference obtained from all imputed data was combined using Rubin's rule; Test type: Superiority — Testing according to the hierarchical testing procedure (only performed if previous outcome measures were statistically significant); p < 0.0001, ANCOVA — Threshold for significance at 0.05 level; LS mean difference = -2.44, 95% CI 2-sided [-2.87 to -2.02]

5. Secondary Outcome: Change From Baseline at Week 24 in the University of Pennsylvania Smell Identification Test (UPSIT) Score
Description: The UPSIT was a 40-item test to measure the individual's ability to detect odors. Total score ranges from 0 (anosmia) to 40 (normal sense of smell), lower score indicated severe smell loss. LS means and SE were obtained from ANCOVA model described in Statistical Analysis Overview. All participants randomized to receive Dupilumab had been on 300 mg q2w regimen until Week 24 and analyzed as a pooled population for Week 24 assessments.
Time Frame: Baseline, Week 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab 300 mg (24 Weeks Pooled Arm)
Number analyzed (Participants) | 150 | 287
score on a scale | -0.81 (0.71) | 9.71 (0.56)
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 300 mg (24 Weeks Pooled Arm); [analysis description as in outcome 4, analysis 1]; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p < 0.0001, ANCOVA — Threshold for significance at 0.05 level; LS mean difference = 10.52, 95% CI 2-sided [8.98 to 12.07]

6. Secondary Outcome: Change From Baseline at Week 24 in Severity of Decreased/Loss of Smell as Assessed by Participant Daily
Description: The severity of decreased/loss of sense of smell was reported by the participants using a 0 to 3 categorical scale (where 0 = no symptoms, 1 = mild symptoms, 2 = moderate symptoms and 3 = severe symptoms), higher score indicated more severe symptoms. LS means and SE were obtained from ANCOVA model described in Statistical Analysis Overview. All participants randomized to receive Dupilumab had been on 300 mg q2w regimen until Week 24 and analyzed as a pooled population for Week 24 assessments.
Time Frame: Baseline, Week 24
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab 300 mg (24 Weeks Pooled Arm)
Number analyzed (Participants) | 153 | 295
score on a scale | -0.23 (0.08) | -1.21 (0.06)
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 300 mg (24 Weeks Pooled Arm); [analysis description as in outcome 4, analysis 1]; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p < 0.0001, ANCOVA — Threshold for significance at 0.05 level; LS mean difference = -0.98, 95% CI 2-sided [-1.15 to -0.81]

7. Secondary Outcome: Change From Baseline at Week 24 in 22-item Sino-nasal Outcome Test (SNOT-22) Scores
Description: The SNOT-22 is a validated questionnaire was used to assess the impact of chronic rhinosinusitis phenotype with nasal polyps (CRSwNP) on health-related quality of life (HRQoL). It is a 22 item questionnaire with each item assigned a score ranging from 0 (no problem) to 5 (problem as bad as it can be). The total score may range from 0 (no disease) to 110 (worst disease), lower scores representing better health related quality of life. LS means and SE were obtained from ANCOVA model described in Statistical Analysis Overview. All participants randomized to receive Dupilumab had been on 300 mg q2w regimen until Week 24 and analyzed as a pooled population for Week 24 assessments.
Time Frame: Baseline, Week 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab 300 mg (24 Weeks Pooled Arm)
Number analyzed (Participants) | 152 | 292
score on a scale | -10.40 (1.61) | -27.77 (1.26)
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 300 mg (24 Weeks Pooled Arm); [analysis description as in outcome 4, analysis 1]; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p < 0.0001, ANCOVA — Threshold for significance at 0.05 level; LS mean difference = -17.36, 95% CI 2-sided [-20.87 to -13.85]

8. Secondary Outcome: Change From Baseline at Week 52 in Nasal Polyp Score
Description: NPS was the sum of right and left nostril scores, as evaluated by means of nasal endoscopy. For each nostril, NPS was graded based on polyp size from 0 to 4 (0 = no polyps to 4 = large polyps causing complete obstruction of the inferior nasal cavity), with a lower score indicating smaller-sized polyps. Total NPS was the sum of right and left nostril scores and ranges from 0 (no polyp) to 8 (large polyp), with highest score representing more severe disease. NPS was assessed by centralized, blinded, independent review of the nasal endoscopy video recordings. Data were analyzed using a hybrid method of the WOCF and MI. LS means and SE were obtained from ANCOVA model described in Statistical Analysis Overview.
Time Frame: Baseline, Week 52
Population: Analysis was performed on ITT population. Here, "overall number of participants analyzed"= participants evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab 300 mg q2w Then q4w | Dupilumab 300 mg q2w
Number analyzed (Participants) | 152 | 145 | 149
score on a scale | 0.16 (0.15) | -2.05 (0.15) | -2.24 (0.15)
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 300 mg q2w Then q4w; [analysis description as in outcome 3, analysis 1]; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p < 0.0001, ANCOVA — Threshold for significance at 0.05 level; LS mean difference = -2.21, 95% CI 2-sided [-2.59 to -1.83] — Dupilumab 300 mg q2w then q4w vs. Placebo
Statistical Analysis 2: Comparison: Placebo vs Dupilumab 300 mg q2w; [analysis description as in outcome 3, analysis 1]; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p < 0.0001, ANCOVA — Threshold for significance at 0.05 level; LS mean difference = -2.41, 95% CI 2-sided [-2.78 to -2.03] — Dupilumab 300 mg q2w vs. Placebo

9. Secondary Outcome: Change From Baseline at Week 52 in Nasal Congestion/Obstruction Symptom Severity Score
Description: NC symptom severity was assessed by the participants on a daily basis from Visit 1 and throughout the study using an e-diary on a scale of 0 to 3, where 0 = no symptoms, 1 = mild symptoms, 2 = moderate symptoms and 3 = severe symptoms, with higher scores indicated more severity. LS means and SE were obtained from ANCOVA model described in Statistical Analysis Overview.
Time Frame: Baseline, Week 52
Population: Analysis was performed on ITT population.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab 300 mg q2w Then q4w | Dupilumab 300 mg q2w
Number analyzed (Participants) | 153 | 145 | 150
score on a scale | -0.37 (0.08) | -1.48 (0.08) | -1.36 (0.07)
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 300 mg q2w Then q4w; [analysis description as in outcome 3, analysis 1]; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p < 0.0001, ANCOVA — Threshold for significance at 0.05 level; LS mean difference = -1.11, 95% CI 2-sided [-1.30 to -0.92] — Dupilumab 300 mg q2w then q4w vs. Placebo
Statistical Analysis 2: Comparison: Placebo vs Dupilumab 300 mg q2w; [analysis description as in outcome 3, analysis 1]; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p < 0.0001, ANCOVA — Threshold for significance at 0.05 level; LS mean difference = -0.99, 95% CI 2-sided [-1.18 to -0.80] — Dupilumab 300 mg q2w vs. Placebo

10. Secondary Outcome: Change From Baseline at Week 52 in 22-item Sino-nasal Outcome Test Scores
Description: The SNOT-22 is a validated questionnaire that was used to assess the impact of CRSwNP on HRQoL. It is a 22 item questionnaire with each item assigned a score ranging from 0 (no problem) to 5 (problem as bad as it can be). The total score may range from 0 (no disease) to 110 (worst disease), lower scores representing better health related quality of life. LS means and SE were obtained from ANCOVA model described in Statistical Analysis Overview.
Time Frame: Baseline, Week 52
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab 300 mg q2w Then q4w | Dupilumab 300 mg q2w
Number analyzed (Participants) | 152 | 145 | 147
score on a scale | -9.06 (1.61) | -30.42 (1.65) | -29.79 (1.64)
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 300 mg q2w Then q4w; [analysis description as in outcome 3, analysis 1]; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p < 0.0001, ANCOVA — Threshold for significance at 0.05 level; LS mean difference = -21.36, 95% CI 2-sided [-25.45 to -17.27] — Dupilumab 300 mg q2w then q4w vs. Placebo
Statistical Analysis 2: Comparison: Placebo vs Dupilumab 300 mg q2w; [analysis description as in outcome 3, analysis 1]; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p < 0.0001, ANCOVA — Threshold for significance at 0.05 level; LS mean difference = -20.73, 95% CI 2-sided [-24.81 to -16.65] — Dupilumab 300 mg q2w vs. Placebo

11. Secondary Outcome: Rescue Treatment Use: Estimate of Percentage of Participants With Greater Than or Equal to (>=) 1 Event by Week 52 Obtained Using Kaplan-Meier Method
Description: Rescue treatment was defined as usage of systemic corticosteroids (SCS) or NP surgery (actual or planned) during the treatment period. Rescue treatment included:
  * SCS: betamethasone, deflazacort, dexamethasone, dexamethasone sodium phosphate, hydrocortisone, meprednisone, methylprednisolone, methylprednisolone sodium succinate, prednisolone, prednisolone sodium succinate, prednisone, stelamin, triamcinolone, and triamcinolone acetonide.
  * Sino-nasal surgery for nasal polyps when there was worsening of signs and/or symptoms during the study.
  Estimate of percentage of participants with event by Week 52 was obtained using Kaplan-Meier method.
Time Frame: Baseline up to 52 weeks
Population: Analysis was performed on ITT population. Data for this outcome measure was planned to be collected and analyzed for the pooled population of participants receiving Dupilumab.
Measure: Number (95% Confidence Interval); unit: percentage of participants with event
Groups:
- Dupilumab 300 mg (Pooled Arm): Pooled arm consisted of all participants who either received Dupilumab 300 mg SC injection q2w from Day 1 of Week 0 up to Week 52 or Dupilumab 300 mg SC injection q2w from Day 1 of Week 0 up to Week 24 and then 300 mg q4w until Week 52, added to background therapy of intranasal MFNS at stable dose.
Arm/Group | Placebo | Dupilumab 300 mg (Pooled Arm)
Number analyzed (Participants) | 153 | 295
percentage of participants with event
  SCS treatment | 42.5 [34.5 to 50.2] | 13.1 [9.0 to 18.0]
  NP surgery | 28.3 [21.2 to 35.7] | 5.5 [2.9 to 9.4]

12. Secondary Outcome: Change From Baseline at Week 52 in Total Symptom Score
Description: The TSS was the sum of participant-assessed nasal symptom scores for NC/obstruction, decreased/loss of sense of smell, and rhinorrhea (anterior/posterior nasal discharge), each accessed on 0-3 categorical scale (where 0 = no symptoms, 1 = mild symptoms, 2 = moderate symptoms and 3 = severe symptoms). Total score ranged from 0 (no symptoms) to 9 (severe symptoms). Higher score indicated more severe symptoms. Data was analyzed using a hybrid method of the WOCF and MI. The imputed completed data were analyzed by fitting an ANCOVA model with corresponding baseline value, treatment group, asthma/NSAID-ERD status, prior surgery history, and regions as covariates.
Time Frame: Baseline, Week 52
Population: Analysis was performed on ITT population.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab 300 mg q2w Then q4w | Dupilumab 300 mg q2w
Number analyzed (Participants) | 153 | 145 | 150
score on a scale | -0.93 (0.20) | -4.17 (0.20) | -3.79 (0.20)

13. Secondary Outcome: Change From Baseline at Week 52 in the University of Pennsylvania Smell Identification Test Score
Description: The UPSIT was a 40-item test to measure the individual's ability to detect odors. Total score ranges from 0 (anosmia) to 40 (normal sense of smell), lower score indicated severe smell loss. Data was analyzed using a hybrid method of the WOCF and MI. The imputed completed data were analyzed by fitting an ANCOVA model with corresponding baseline value, treatment group, asthma/NSAID-ERD status, prior surgery history, and regions as covariates.
Time Frame: Baseline, Week 52
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab 300 mg q2w Then q4w | Dupilumab 300 mg q2w
Number analyzed (Participants) | 150 | 142 | 145
score on a scale | -0.78 (0.71) | 9.99 (0.73) | 9.53 (0.72)

14. Secondary Outcome: Change From Baseline at Week 52 in Severity of Decreased/Loss of Smell
Description: The severity of decreased/loss of sense of smell was reported by the participants using a 0 to 3 categorical scale (where 0 = no symptoms, 1 = mild symptoms, 2 = moderate symptoms and 3 = severe symptoms), higher score indicated more severe symptoms. Data was analyzed using a hybrid method of the WOCF and MI. The imputed completed data were analyzed by fitting an ANCOVA model with corresponding baseline value, treatment group, asthma/NSAID-ERD status, prior surgery history, and regions as covariates.
Time Frame: Baseline, Week 52
Population: Analysis was performed on ITT population.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab 300 mg q2w Then q4w | Dupilumab 300 mg q2w
Number analyzed (Participants) | 153 | 145 | 150
score on a scale | -0.18 (0.09) | -1.49 (0.09) | -1.29 (0.08)

15. Secondary Outcome: Change From Baseline at Week 52 in Opacification of Sinuses Measured by Lund-Mackay Score
Description: The LMK scoring system rated each of both the left and right frontal, maxillary, sphenoid, ostiomeatal complex, anterior ethmoid and posterior ethmoid sinuses using following grading: 0 = normal, 1 = partial opacification, 2 = total opacification. The total score was the sum of scores from each side and ranges from 0 (normal) to 24 (more opacified); higher score indicated more severe disease. Data was analyzed using a hybrid method of the WOCF and MI. The imputed completed data were analyzed by fitting an ANCOVA model with corresponding baseline value, treatment group, asthma/NSAID-ERD status, prior surgery history, and regions as covariates.
Time Frame: Baseline, Week 52
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab 300 mg q2w Then q4w | Dupilumab 300 mg q2w
Number analyzed (Participants) | 150 | 140 | 149
score on a scale | 0.11 (0.37) | -5.60 (0.37) | -6.83 (0.37)

16. Secondary Outcome: Change From Baseline at Week 24 in Visual Analogue Scale (VAS) for Rhinosinusitis
Description: The VAS for rhinosinusitis was used to evaluate the total disease severity. The participants were asked to indicate on a 10 centimeters VAS the answer to the question, "How troublesome are your symptoms of your rhinosinusitis?" The range of the VAS was from 0 (not troublesome) to 10 (worse thinkable troublesome), where higher score indicated worse thinkable troublesome. Data was analyzed using a hybrid method of the WOCF and MI. The imputed completed data were analyzed by fitting an ANCOVA model with corresponding baseline value, treatment group, asthma/NSAID-ERD status, prior surgery history, and regions as covariates. All participants randomized to receive Dupilumab had been on 300 mg q2w regimen until Week 24 and analyzed as a pooled population for Week 24 assessments.
Time Frame: Baseline, Week 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: centimeters
Arm/Group | Placebo | Dupilumab 300 mg (24 Weeks Pooled Arm)
Number analyzed (Participants) | 150 | 289
centimeters | -1.39 (0.24) | -4.32 (0.19)

17. Secondary Outcome: Change From Baseline at Week 52 in Visual Analogue Scale for Rhinosinusitis
Description: The VAS for rhinosinusitis was used to evaluate the total disease severity. The participants were asked to indicate on a 10 centimeters VAS the answer to the question, "How troublesome are your symptoms of your rhinosinusitis?" The range of the VAS was from 0 (not troublesome) to 10 (worse thinkable troublesome), where higher score indicated worse thinkable troublesome. Data was analyzed using a hybrid method of the WOCF and MI. The imputed completed data were analyzed by fitting an ANCOVA model with corresponding baseline value, treatment group, asthma/NSAID-ERD status, prior surgery history, and regions as covariates.
Time Frame: Baseline, Week 52
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: centimeters
Arm/Group | Placebo | Dupilumab 300 mg q2w Then q4w | Dupilumab 300 mg q2w
Number analyzed (Participants) | 150 | 143 | 146
centimeters | -0.93 (0.26) | -4.39 (0.26) | -4.74 (0.26)

18. Secondary Outcome: Change From Baseline at Week 24 in Nasal Peak Inspiratory Flow (NPIF)
Description: NPIF evaluation represented a physiologic measure of the air flow through both nasal cavities during forced inspiration expressed in liters per minute. Higher NPIF values were indicative of better nasal air flow. Data was analyzed using a hybrid method of the WOCF and MI. The imputed completed data were analyzed by fitting an ANCOVA model with corresponding baseline value, treatment group, asthma/NSAID-ERD status, prior surgery history, and regions as covariates. All participants randomized to receive Dupilumab had been on 300 mg q2w regimen until Week 24 and analyzed as a pooled population for Week 24 assessments.
Time Frame: Baseline, Week 24
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: liters per minute
Arm/Group | Placebo | Dupilumab 300 mg (24 Weeks Pooled Arm)
Number analyzed (Participants) | 153 | 295
liters per minute | 18.65 (3.95) | 55.29 (3.08)

19. Secondary Outcome: Change From Baseline at Week 24 in Rhinorrhea Daily Symptom Score
Description: Rhinorrhea was reported by the participants using a 0 to 3 categorical scale (where 0 = no symptoms, 1 = mild symptoms, 2 = moderate symptoms and 3 = severe symptoms), where higher scores indicated more severe symptoms. Data was analyzed using a hybrid method of the WOCF and MI. The imputed completed data were analyzed by fitting an ANCOVA model with corresponding baseline value, treatment group, asthma/NSAID-ERD status, prior surgery history, and regions as covariates. All participants randomized to receive Dupilumab had been on 300 mg q2w regimen until Week 24 and analyzed as a pooled population for Week 24 assessments.
Time Frame: Baseline, Week 24
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab 300 mg (24 Weeks Pooled Arm)
Number analyzed (Participants) | 153 | 295
score on a scale | -0.40 (0.07) | -0.99 (0.05)

20. Secondary Outcome: Change From Baseline at Week 52 in Rhinorrhea Daily Symptom Score
Description: Rhinorrhea was reported by the participants using a 0 to 3 categorical scale (where 0 = no symptoms, 1 = mild symptoms, 2 = moderate symptoms and 3 = severe symptoms), where higher scores indicated more severe symptoms. Data was analyzed using a hybrid method of the WOCF and MI. The imputed completed data were analyzed by fitting an ANCOVA model with corresponding baseline value, treatment group, asthma/NSAID-ERD status, prior surgery history, and regions as covariates.
Time Frame: Baseline, Week 52
Population: Analysis was performed on ITT population.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab 300 mg q2w Then q4w | Dupilumab 300 mg q2w
Number analyzed (Participants) | 153 | 145 | 150
score on a scale | -0.35 (0.07) | -1.19 (0.07) | -1.15 (0.07)

21. Secondary Outcome: Mean Total Systemic Corticosteroids Rescue Dose Prescribed During Treatment Period
Description: SCS included: betamethasone, deflazacort, dexamethasone, dexamethasone sodium phosphate, hydrocortisone, meprednisone, methylprednisolone, methylprednisolone sodium succinate, prednisolone, prednisolone sodium succinate, prednisone, stelamin, triamcinolone, and triamcinolone acetonide. For every participant, the total dose was calculated as (prescribed total daily dose*duration of SCS use). Then, mean of the total dose of 64 participants (placebo group), 17 participants (dupilumab 300 mg q2w then q4w) and 22 participants (dupilumab 300 mg q2w) was derived.
Time Frame: Baseline to Week 52
Population: The analysis was performed on ITT population. Here, "overall number of participants analyzed" signifies participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | Placebo | Dupilumab 300 mg q2w Then q4w | Dupilumab 300 mg q2w
Number analyzed (Participants) | 64 | 17 | 22
milligrams | 547.56 (665.40) | 282.38 (243.15) | 389.68 (502.61)

22. Secondary Outcome: Total Systemic Corticosteroids Rescue Intake Duration: Average Duration Per Participant
Description: Rescue treatment was defined as usage of SCS or NP surgery (actual or planned) during the treatment period. SCS Rescue intake duration was defined as the duration (in days) from start of SCS rescue medication till the end of SCS rescue treatment.
Time Frame: Baseline to Week 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Placebo | Dupilumab 300 mg q2w Then q4w | Dupilumab 300 mg q2w
Number analyzed (Participants) | 64 | 17 | 22
days | 19.58 (17.67) | 10.71 (9.00) | 23.23 (55.23)

23. Secondary Outcome: Changed From Baseline at Week 24 in Forced Expiratory Volume in 1 Second (FEV1) for Participants With Asthma
Description: FEV1 was the volume of air exhaled in the first second of a forced expiration as measured by spirometer. Data was analyzed using a hybrid method of the WOCF and MI. The imputed completed data were analyzed by fitting an ANCOVA model with corresponding baseline value, treatment group, prior surgery history, and regions as covariates. All participants randomized to receive Dupilumab had been on 300 mg q2w regimen until Week 24 and analyzed as a pooled population for Week 24 assessments.
Time Frame: Baseline, Week 24
Population: Analysis was performed on a subset of participants which included all randomized participants with asthma and had available data for this outcome measure. Data for this outcome measure was planned to be analyzed for the combined population of participants who received Dupilumab.
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo | Dupilumab 300 mg (24 Weeks Pooled Arm)
Number analyzed (Participants) | 90 | 176
liters | -0.05 (0.05) | 0.17 (0.04)

24. Secondary Outcome: Change From Baseline at Week 52 in Forced Expiratory Volume in 1 Second for Participants With Asthma
Description: FEV1 was the volume of air exhaled in the first second of a forced expiration as measured by spirometer. Data was analyzed using a hybrid method of the WOCF and MI. The imputed completed data were analyzed by fitting an ANCOVA model with corresponding baseline value, treatment group, prior surgery history, and regions as covariates.
Time Frame: Baseline, Week 52
Population: Analysis was performed on a subset of participants which included all randomized participants with asthma and had available data for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo | Dupilumab 300 mg q2w Then q4w | Dupilumab 300 mg q2w
Number analyzed (Participants) | 90 | 91 | 85
liters | -0.18 (0.05) | 0.10 (0.05) | 0.06 (0.05)

25. Secondary Outcome: Change From Baseline at Week 24 in Asthma Control Questionnaire-6 (ACQ-6) for Participants With Asthma
Description: ACQ-6 had 6 questions which assessed the most common asthma symptoms (woken by asthma, symptoms on waking, activity limitation, shortness of breath, wheezing, puffs/inhalations use). Participants were asked to recall how their asthma had been during the previous week and to respond to the symptom questions on a 7-point scale ranged from 0 = no impairment to 6 = maximum impairment. The ACQ-6 score was the mean of the scores of all 6 questions and therefore, ranged from 0 (totally controlled) to 6 (severely uncontrolled), with higher scores indicated lower asthma control. Data were analyzed using a hybrid method of the WOCF and MI. The imputed completed data were analyzed by fitting an ANCOVA model with corresponding baseline value, treatment, asthma status, prior surgery history, and regions as covariates. All participants randomized to receive Dupilumab had been on 300 mg q2w regimen until Week 24 and analyzed as a pooled population for Week 24 assessments.
Time Frame: Baseline, Week 24
Population: as for outcome 23
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab 300 mg (24 Weeks Pooled Arm)
Number analyzed (Participants) | 90 | 171
score on a scale | 0.08 (0.09) | -0.78 (0.07)

26. Secondary Outcome: Change From Baseline at Week 52 in Asthma Control Questionnaire-6 for Participants With Asthma
Description: ACQ-6 had 6 questions which assessed the most common asthma symptoms (woken by asthma, symptoms on waking, activity limitation, shortness of breath, wheezing, puffs/inhalations use). Participants were asked to recall how their asthma had been during the previous week and to respond to the symptom questions on a 7-point scale ranged from 0 = no impairment to 6 = maximum impairment. The ACQ-6 score was the mean of the scores of all 6 questions and therefore, ranged from 0 (totally controlled) to 6 (severely uncontrolled), with higher scores indicated lower asthma control. Data were analyzed using a hybrid method of the WOCF and MI. The imputed completed data were analyzed by fitting an ANCOVA model with corresponding baseline value, treatment, asthma status, prior surgery history, and regions as covariates.
Time Frame: Baseline, Week 52
Population: as for outcome 24
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab 300 mg q2w Then q4w | Dupilumab 300 mg q2w
Number analyzed (Participants) | 90 | 89 | 82
score on a scale | 0.12 (0.10) | -0.76 (0.10) | -0.83 (0.10)

27. Secondary Outcome: Change From Baseline at Week 24 in Nasal Congestion/Obstruction Symptom Severity Score: Subgroup of Participants With Asthma
Description: NC symptom severity was assessed by the participants on a daily basis from Visit 1 and throughout the study using an e-diary on a scale of 0 to 3, where 0 = no symptoms, 1 = mild symptoms, 2 = moderate symptoms and 3 = severe symptoms, with higher scores indicated more severity. Data were analyzed using a hybrid method of the WOCF and MI. The imputed completed data were analyzed by fitting ANCOVA model with corresponding baseline, treatment group, prior surgery history, and regions as covariates. All participants randomized to receive Dupilumab had been on 300 mg q2w regimen until Week 24 and analyzed as a pooled population for Week 24 assessments.
Time Frame: Baseline, Week 24
Population: Analysis was performed on a subset of participants which included all randomized participants with asthma.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab 300 mg (24 Weeks Pooled Arm)
Number analyzed (Participants) | 91 | 176
score on a scale | -0.39 (0.09) | -1.36 (0.07)

28. Secondary Outcome: Change From Baseline at Week 52 in Nasal Congestion/Obstruction Symptom Severity Score: Subgroup of Participants With Asthma
Description: NC symptom severity was assessed by the participants on a daily basis from Visit 1 and throughout the study using an e-diary on a scale of 0 to 3, where 0 = no symptoms, 1 = mild symptoms, 2 = moderate symptoms and 3 = severe symptoms, with higher scores indicated more severity. Data were analyzed using a hybrid method of the WOCF and MI. The imputed completed data were analyzed by fitting ANCOVA model with corresponding baseline, treatment group, prior surgery history, and regions as covariates.
Time Frame: Baseline, Week 52
Population: Analysis was performed on a subset of participants which included all randomized participants with asthma.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab 300 mg q2w Then q4w | Dupilumab 300 mg q2w
Number analyzed (Participants) | 91 | 91 | 85
score on a scale | -0.34 (0.09) | -1.51 (0.09) | -1.44 (0.09)

29. Secondary Outcome: Change From Baseline at Week 24 in Nasal Congestion/Obstruction Symptom Severity Score: Subgroup of Participants With Prior Nasal Polyp Surgery
Description: as for outcome 27
Time Frame: Baseline, Week 24
Population: Analysis was performed on a subset of participants which included all randomized participants with prior NP surgery history.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab 300 mg (24 Weeks Pooled Arm)
Number analyzed (Participants) | 88 | 173
score on a scale | -0.27 (0.10) | -1.30 (0.08)

30. Secondary Outcome: Change From Baseline at Week 52 in Nasal Congestion/Obstruction Symptom Severity Score: Subgroup of Participants With Prior Nasal Polyp Surgery
Description: NC symptom severity was assessed by the participants on a daily basis from Visit 1 and throughout the study using an e-diary on a scale of 0 to 3, where 0 = no symptoms, 1 = mild symptoms, 2 = moderate symptoms and 3 = severe symptoms, with higher scores indicated more severity. Data were analyzed using a hybrid method of the WOCF and MI. The imputed completed data were analyzed by fitting an ANCOVA model with corresponding baseline, treatment group, asthma/NSAID-ERD status, and regions as covariates.
Time Frame: Baseline, Week 52
Population: as for outcome 29
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab 300 mg q2w Then q4w | Dupilumab 300 mg q2w
Number analyzed (Participants) | 88 | 85 | 88
score on a scale | -0.25 (0.10) | -1.54 (0.10) | -1.35 (0.09)

31. Secondary Outcome: Change From Baseline at Week 24 in Nasal Polyp Score: Subgroup of Participants With Asthma
Description: NPS was the sum of right and left nostril scores, as evaluated by means of nasal endoscopy. For each nostril, NPS was graded from 0 to 4 (0 = no polyps to 4 = large polyps causing complete obstruction of the inferior nasal cavity), with a lower score indicating smaller-sized polyps. Total NPS was the sum of right and left nostril scores and ranges from 0 (no polyp) to 8 (large polyp), with highest score representing more severe disease. NPS was assessed by centralized, blinded, independent review of the nasal endoscopy video recordings. Data were analyzed using a hybrid method of the WOCF and MI. LS mean and SE were obtained from ANCOVA model. All participants randomized to receive Dupilumab had been on 300 mg q2w regimen until Week 24 and analyzed as a pooled population for Week 24 assessments.
Time Frame: Baseline, Week 24
Population: as for outcome 24
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab 300 mg (24 Weeks Pooled Arm)
Number analyzed (Participants) | 90 | 176
score on a scale | 0.13 (0.17) | -1.88 (0.13)

32. Secondary Outcome: Change From Baseline at Week 52 in Nasal Polyp Score: Subgroup of Participants With Asthma
Description: NPS was the sum of right and left nostril scores, as evaluated by means of nasal endoscopy. For each nostril, NPS was graded from 0 to 4 (0 = no polyps to 4 = large polyps causing complete obstruction of the inferior nasal cavity), with a lower score indicating smaller-sized polyps. Total NPS was the sum of right and left nostril scores and ranges from 0 (no polyp) to 8 (large polyp), with highest score representing more severe disease. NPS was assessed by centralized, blinded, independent review of the nasal endoscopy video recordings. Data were analyzed using a hybrid method of the WOCF and MI. LS mean and SE were obtained from ANCOVA model.
Time Frame: Baseline, Week 52
Population: as for outcome 24
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab 300 mg q2w Then q4w | Dupilumab 300 mg q2w
Number analyzed (Participants) | 90 | 91 | 85
score on a scale | 0.29 (0.20) | -2.25 (0.20) | -2.34 (0.20)

33. Secondary Outcome: Change From Baseline at Week 24 in Nasal Polyp Score: Subgroup of Participants With Prior Nasal Polyp Surgery
Description: as for outcome 31
Time Frame: Baseline, Week 24
Population: Analysis was performed on a subset of participants which included all randomized participants with prior NP surgery history and had available data for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab 300 mg (24 Weeks Pooled Arm)
Number analyzed (Participants) | 88 | 172
score on a scale | 0.22 (0.19) | -1.73 (0.15)

34. Secondary Outcome: Change From Baseline at Week 52 in Nasal Polyp Score: Subgroup of Participants With Prior Nasal Polyp Surgery
Description: as for outcome 32
Time Frame: Baseline, Week 52
Population: as for outcome 33
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab 300 mg q2w Then q4w | Dupilumab 300 mg q2w
Number analyzed (Participants) | 88 | 85 | 87
score on a scale | 0.21 (0.21) | -2.22 (0.22) | -2.56 (0.21)

35. Secondary Outcome: Change From Baseline at Week 24 in Opacification of Sinuses Measured by Lund Mackay Score: Subgroup of Participants With Asthma
Description: The LMK scoring system rated each of both the left and right frontal, maxillary, sphenoid, ostiomeatal complex, anterior ethmoid and posterior ethmoid sinuses using following grading: 0 = normal, 1 = partial opacification, 2 = total opacification. The total score was the sum of scores from each side and ranges from 0 (normal) to 24 (more opacified); higher score indicated more severe disease. Data was analyzed using a hybrid method of the WOCF and MI. The imputed completed data were analyzed by fitting an ANCOVA model with corresponding baseline value, treatment group, asthma/NSAID-ERD status, prior surgery history, and regions as covariates. All participants randomized to receive Dupilumab had been on 300 mg q2w regimen until Week 24 and analyzed as a pooled population for Week 24 assessments.
Time Frame: Baseline, Week 24
Population: as for outcome 24
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab 300 mg (24 Weeks Pooled Arm)
Number analyzed (Participants) | 89 | 174
score on a scale | -0.33 (0.40) | -5.86 (0.31)

36. Secondary Outcome: Change From Baseline at Week 52 in Opacification of Sinuses Measured by Lund Mackay Score: Subgroup of Participants With Asthma
Description: as for outcome 15
Time Frame: Baseline, Week 52
Population: as for outcome 24
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab 300 mg q2w Then q4w | Dupilumab 300 mg q2w
Number analyzed (Participants) | 89 | 89 | 85
score on a scale | -0.20 (0.46) | -6.23 (0.45) | -7.22 (0.47)

37. Secondary Outcome: Change From Baseline at Week 24 in Opacification of Sinuses Measured by Lund Mackay Score: Subgroup of Participants With Prior Nasal Polyp Surgery
Description: The LMK scoring system rated each of both the left and right frontal, maxillary, sphenoid, ostiomeatal complex, anterior ethmoid and posterior ethmoid sinuses using following grading: 0 = normal, 1 = partial opacification, 2 = total opacification. The total score was the sum of scores from each side and ranges from 0 (normal) to 24 (more opacified); higher score indicated more severe disease. Data were analyzed using a hybrid method of the WOCF and MI. The imputed completed data were analyzed by fitting an ANCOVA model with corresponding baseline, treatment group, asthma/NSAID-ERD status, and regions as covariates. All participants randomized to receive Dupilumab had been on 300 mg q2w regimen until Week 24 and analyzed as a pooled population for Week 24 assessments.
Time Frame: Baseline, Week 24
Population: as for outcome 33
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab 300 mg (24 Weeks Pooled Arm)
Number analyzed (Participants) | 85 | 169
score on a scale | -0.10 (0.42) | -5.42 (0.33)

38. Secondary Outcome: Change From Baseline at Week 52 in Opacification of Sinuses Measured by Lund Mackay Score: Subgroup of Participants With Prior Nasal Polyp Surgery
Description: The LMK scoring system rated each of both the left and right frontal, maxillary, sphenoid, ostiomeatal complex, anterior ethmoid and posterior ethmoid sinuses using following grading: 0 = normal, 1 = partial opacification, 2 = total opacification. The total score was the sum of scores from each side and ranges from 0 (normal) to 24 (more opacified); higher score indicated more severe disease. Data were analyzed using a hybrid method of the WOCF and MI. The imputed completed data were analyzed by fitting an ANCOVA model with corresponding baseline, treatment group, asthma/NSAID-ERD status, and regions as covariates.
Time Frame: Baseline, Week 52
Population: as for outcome 33
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab 300 mg q2w Then q4w | Dupilumab 300 mg q2w
Number analyzed (Participants) | 85 | 82 | 87
score on a scale | -0.06 (0.50) | -6.01 (0.50) | -7.45 (0.49)

39. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs) and TEAEs Leading to Treatment Discontinuation
Description: An Adverse Event (AE) was defined as any untoward medical occurrence that did not necessarily have to have a causal relationship with the study treatment. TEAEs were defined as AEs that developed or worsened in grade or became serious during TEAE period which was defined as the period from the time of first dose of drug until 84 days following the last administration of drug. SAE was defined as any untoward medical occurrence that at any dose: results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is a medically important event.
Time Frame: Baseline up to 84 days after last dose of study drug (up to 64 weeks)
Population: Analysis was performed on safety population which included all participants who received at least 1 dose or part of a dose of the investigational medicinal product (IMP), analyzed according to the treatment actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Dupilumab 300 mg q2w Then q4w | Dupilumab 300 mg q2w
Number analyzed (Participants) | 150 | 148 | 149
Participants
  Any TEAE | 138 | 134 | 125
  Any treatment emergent SAE | 16 | 12 | 8
  Any TEAE leading to death | 0 | 1 | 0
  TEAE leading to treatment discontinuation | 17 | 2 | 6

40. Secondary Outcome: Change From Baseline at Week 24 in European Quality of Life 5 Dimension Scale (EQ-5D) Visual Analog Scale Score
Description: The EQ-5D was a standardized HRQoL questionnaire consisting of EQ-5D descriptive system and EQ VAS. The EQ-5D descriptive system comprised of 5 dimensions: mobility, selfcare, usual activities, pain/discomfort and anxiety/depression. Each dimension had 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. EQ VAS recorded the participant's self-rated health on a vertical VAS that allowed them to indicate their health state that can range from 0 (worst imaginable) to 100 (best imaginable). All participants randomized to receive Dupilumab had been on 300 mg q2w regimen until Week 24 and analyzed as a pooled population for Week 24 assessments.
Time Frame: Baseline, Week 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab 300 mg (24 Weeks Pooled Arm)
Number analyzed (Participants) | 151 | 289
score on a scale | 3.91 (1.50) | 10.83 (1.16)

41. Secondary Outcome: Change From Baseline at Week 52 in European Quality of Life 5 Dimension Scale Visual Analog Scale Score
Description: The EQ-5D was a standardized HRQoL questionnaire consisting of EQ-5D descriptive system and EQ VAS. The EQ-5D descriptive system comprised of 5 dimensions: mobility, selfcare, usual activities, pain/discomfort and anxiety/depression. Each dimension had 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. EQ VAS recorded the participant's self-rated health on a vertical VAS that allowed them to indicate their health state that can range from 0 (worst imaginable) to 100 (best imaginable).
Time Frame: Baseline, Week 52
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab 300 mg q2w Then q4w | Dupilumab 300 mg q2w
Number analyzed (Participants) | 151 | 143 | 146
score on a scale | 1.38 (1.60) | 11.98 (1.63) | 13.14 (1.62)

42. Secondary Outcome: Functional Dupilumab Concentration in Serum
Time Frame: Baseline, Week 2, Week 4, Week 16, Week 24, Week 40, End of treatment (Week 52), End of study (Week 64)
Population: Analysis performed on pharmacokinetics population (PK) which included all participants who received at least 1 dose of IMP with at least 1 evaluable functional dupilumab concentration result. Here, 'number analyzed' = number of participants with available data for each time point. PK data was not collected and assessed for the placebo arm.
Measure: Mean (Standard Deviation); unit: nanogram/milliliter
Groups:
- Dupilumab 300 mg q2w Then q4w: Dupilumab 300 mg SC injection q2w from Day 1 of Week 0 up to Week 24 and then 300 mg q4w until Week 52 added to background therapy of intranasal MFNS at stable dose. After Week 24, Dupilumab administration was alternated with matched placebo injection every other week up to Week 50. One participant randomized to dupilumab 300 mg q2w arm received 1 dose of placebo and was counted in the 300 mg q2w then q4w arm.
Arm/Group | Dupilumab 300 mg q2w Then q4w | Dupilumab 300 mg q2w
Number analyzed (Participants) | 146 | 149
nanogram/milliliter
  Baseline: number analyzed (Participants) | 145 | 146
  Baseline | 0.00 (0.00) | 0.00 (0.00)
  Week 2: number analyzed (Participants) | 143 | 146
  Week 2 | 21545.79 (9120.36) | 22285.67 (8459.01)
  Week 4: number analyzed (Participants) | 144 | 144
  Week 4 | 33760.62 (16419.72) | 37326.31 (14226.12)
  Week 16: number analyzed (Participants) | 143 | 141
  Week 16 | 70503.07 (31234.86) | 74382.04 (33118.68)
  Week 24: number analyzed (Participants) | 144 | 143
  Week 24 | 75929.41 (35466.00) | 79890.06 (35361.97)
  Week 40: number analyzed (Participants) | 141 | 138
  Week 40 | 21052.06 (18588.68) | 80526.37 (34048.41)
  Week 52: number analyzed (Participants) | 141 | 135
  Week 52 | 17276.13 (16353.20) | 75872.58 (34127.85)
  Week 64: number analyzed (Participants) | 139 | 135
  Week 64 | 53.60 (160.53) | 851.30 (2682.21)

43. Secondary Outcome: Number of Participants With Treatment-Emergent And Treatment-Boosted Anti-drug Antibodies Response (ADA)
Description: ADA response were categorized as: treatment emergent and treatment boosted response. 1) Treatment emergent was defined as a positive response in the ADA assay post first dose, when baseline results are negative or missing. 2) Treatment boosted was defined as: an ADA positive response in the assay post first dose that is greater-than or equal to 4-fold over baseline titer levels, when baseline results are positive.
Time Frame: Baseline to Week 52
Population: The analysis was performed on ADA population which included participants who received at least 1 dose of IMP with at least one evaluable ADA serum sample that was assayed successfully in the ADA assay (either 'ADA negative' or 'ADA positive') following the first dose of the study medication.
Measure: Count of Participants; unit: Participants
Groups:
- Dupilumab 300 mg q2w Then q4w: Dupilumab 300 mg SC injection q2w from Day 1 of Week 0 up to Week 24 and then 300 mg q4w until Week 52 added to background therapy of intranasal MFNS at stable dose. After Week 24, Dupilumab administration was alternated with matched placebo injection every other week up to Week 50. Two participants randomized to placebo arm accidently received 1 dose of dupilumab 300 mg and counted in the 300 mg q2w then q4w arm. One participant randomized to the dupilumab 300 mg q2w arm received 1 dose of placebo and was counted in the 300 mg q2w then q4w arm.
Arm/Group | Placebo | Dupilumab 300 mg q2w Then q4w | Dupilumab 300 mg q2w
Number analyzed (Participants) | 149 | 148 | 148
Participants
  With treatment-emergent ADA | 6 | 18 | 8
  With treatment-boosted ADA | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) were collected from signature of the informed consent form up to 64 weeks regardless of seriousness or relationship to investigational product.
Description: Reported AEs are treatment emergent AEs that developed/worsened during the 'on treatment period' (defined as the period from the time of first dose of drug until 84 days following the last administration of drug). Analysis was performed on safety population.
Arm/Group | Placebo | Dupilumab 300 mg q2w Then q4w | Dupilumab 300 mg q2w
All-Cause Mortality (participants affected / at risk) | 0/150 | 1/148 | 0/149
Serious Adverse Events (participants affected / at risk) | 16/150 | 12/148 | 8/149
Other Adverse Events (participants affected / at risk) | 111/150 | 95/148 | 90/149
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=150) | Dupilumab 300 mg q2w Then q4w (N=148) | Dupilumab 300 mg q2w (N=149)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Deafness Neurosensory (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Vestibular Disorder (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Retinal Vein Thrombosis (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal Angiectasia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oesophageal Perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Eosinophilic Granulomatosis With Polyangiitis (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Chronic Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Corneal Abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infectious Pleural Effusion (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Septic Shock (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Wound Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Facial Bones Fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Femur Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Hand Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Humerus Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Open Globe Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Traumatic Intracranial Haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Upper Limb Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Weight Decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Nasal Neoplasm Benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Temporal Lobe Epilepsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Asthmatic Crisis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Chronic Rhinosinusitis With Nasal Polyps (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nasal Polyps (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 0 (0)
Miscarriage Of Partner (Social circumstances) | 1 (1) | 0 (0) | 0 (0)
Peripheral Arterial Occlusive Disease (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=150) | Dupilumab 300 mg q2w Then q4w (N=148) | Dupilumab 300 mg q2w (N=149)
Injection Site Erythema (General disorders) | 11 (28) | 10 (26) | 11 (25)
Injection Site Reaction (General disorders) | 3 (4) | 8 (24) | 5 (15)
Acute Sinusitis (Infections and infestations) | 16 (18) | 5 (5) | 5 (8)
Bronchitis (Infections and infestations) | 8 (13) | 9 (10) | 9 (10)
Nasopharyngitis (Infections and infestations) | 38 (48) | 31 (53) | 33 (50)
Sinusitis (Infections and infestations) | 17 (29) | 14 (19) | 9 (9)
Upper Respiratory Tract Infection (Infections and infestations) | 20 (23) | 8 (9) | 10 (13)
Accidental Overdose (Injury, poisoning and procedural complications) | 11 (12) | 12 (13) | 5 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 12 (12) | 7 (9)
Back Pain (Musculoskeletal and connective tissue disorders) | 10 (11) | 5 (6) | 8 (11)
Headache (Nervous system disorders) | 18 (31) | 17 (32) | 14 (17)
Asthma (Respiratory, thoracic and mediastinal disorders) | 20 (31) | 15 (23) | 8 (11)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (11) | 9 (10) | 9 (13)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 20 (22) | 8 (10) | 13 (16)
Nasal Polyps (Respiratory, thoracic and mediastinal disorders) | 26 (51) | 20 (20) | 9 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2017-05-17): https://cdn.clinicaltrials.gov/large-docs/54/NCT02898454/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-14): https://cdn.clinicaltrials.gov/large-docs/54/NCT02898454/SAP_001.pdf